CLINICAL TRIAL: NCT03812965
Title: Effectiveness and Durability of Botulinum Toxin Application in the Treatment of Gingival Smile
Brief Title: Botulinum Toxin in the Treatment of Gingival Smile
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Ibirapuera (Other)
Responsible Party: Principal Investigator, Karen Müller Ramalho, Full Professor, Universidade Ibirapuera
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 80103617.0.0000.5597
Record Dates: First submitted 2019-01-17; First posted 2019-01-23 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Smiling
Keywords: Botulinum Toxin; Gingival Smile
MeSH Terms: conditions — Smiling | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Botulinum Toxin type A (4 points of application) (Experimental): 4 points of Botulinum Toxin application in the muscles: Levators labii superioris alaeque nasi muscle and Levators labii superioris muscle (n=10 Patients)
  Interventions: Drug: Botulinum toxin type A
- Group 2 - - Botulinum Toxin type A (2 points of application) (Experimental): 2 points of Botulinum Toxin application in the muscles: Levators labii superioris alaeque nasi muscle (n=10 Patients)
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — 2 units/point of botulinum toxin type A

SUMMARY:
Objective: to evaluate the effect of two gingival smile treatment techniques using botulinum toxin. Materials and methods: The randomized, double-blind clinical trial (patient and examiner) will be conducted by two trained and calibrated dentists. Ten patients will be randomly assigned to each group, in a total of 20 patients with gingiva smile greater than or equal to 3mm. In group 1, 10 patients will receive 2 units/point of botulinum toxin Botulift® (botulinum toxin type A), in the muscles form the face: Levators labii superioris alaeque nasi muscle and Levators labii superioris muscle, totalizing 4 points. In group 2, 2 units/point was injected in the muscles: levators labii superioris alaeque nasi muscle, totalizing 2 points. The amount of exposed gingiva during smile will be measured using a pachymeter and the muscle activity of the region will be evaluated through electromyography, before and after treatment (2, 8, 12, 21 and 25 weeks). Patient satisfaction and discomfort due to treatment will be evaluated in the same periods through questionnaire. The impact of the treatment in life quality will be evaluated through OHIP-14 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders exhibiting gingival exposure greater than or equal to 3 mm above the central incisor during smile
2. Patients with good general health and good oral hygiene.

Exclusion Criteria:

1. Patients with Botulinum Toxin allergy or albumin, or who have previously performed botulinum toxin facial treatment previously.
2. Patients with Amyotrophic Lateral Sclerosis, Neuropathy, Myasthenia Gravis or Lambert-Eaton Syndrome, women who are pregnant or planning to become pregnant, are breastfeeding women.
3. Patients who are participating in other research involving other drugs.
4. Patients who use drugs that interfere with neuromuscular transmission

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Exposed Gingiva during Smile (mm) | Before Treatment
  Measurement of exposed gingiva during smile using a pachymeter
Exposed Gingiva during Smile (mm) | After Treatment (2 weeks)
  Measurement of exposed gingiva during smile using a pachymeter
Exposed Gingiva during Smile (mm) | After Treatment (8 weeks)
  Measurement of exposed gingiva during smile using a pachymeter
Exposed Gingiva during Smile (mm) | After Treatment (12 weeks)
  Measurement of exposed gingiva during smile using a pachymeter
Exposed Gingiva during Smile (mm) | After Treatment (21 weeks)
  Measurement of exposed gingiva during smile using a pachymeter
Exposed Gingiva during Smile (mm) | After Treatment (25 weeks)
  Measurement of exposed gingiva during smile using a pachymeter

SECONDARY OUTCOMES:
Muscles Activity | Before Treatment
  Muscles activity using electromyography
Muscles Activity | After Treatment (2 weeks)
  Muscles activity using electromyography
Muscles Activity | After Treatment (8 weeks)
  Muscles activity using electromyography
Muscles Activity | After Treatment (12 weeks)
  Muscles activity using electromyography
Muscles Activity | After Treatment (21 weeks)
  Muscles activity using electromyography
Muscles Activity | After Treatment (25 weeks)
  Muscles activity using electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Aline B Costa, DDS, Study Chair — Ibirapuera University; Dinete Romansina, MSc, Study Chair — University of Sao Paulo; Juliana Ramalho, DDS, Study Chair — Ibirapuera University; Karen M Ramalho, PhD, Principal Investigator — Ibirapuera University; Susana Morimoto, PhD, Study Chair — Ibirapuera University
Locations (1):
- Universidade Ibirapuera, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided